CLINICAL TRIAL: NCT04801355
Title: Single-center, Randomized Trial: Full-thickness Laparo-endoscopic Excision vs Laparoscopic Colectomy for Colonic Tumors
Brief Title: Full-thickness Laparo-endoscopic Excision vs Laparoscopic Colectomy for Colonic Tumors
Acronym: FlexLaC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Achkasov Sergey, Head of colorectal surgery and oncology department, State Scientific Centre of Coloproctology, Russian Federation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201
Record Dates: First submitted 2021-03-08; First posted 2021-03-17 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Neoplasms, Benign
Keywords: Full-thickness laparo-endoscopic; Colorectal tumors; Laparoscopic resection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Laparo-endoscopic full-thickness colon resection
Who Masked: Participant, Investigator
Masking Description: patients with colon adenomas
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic resection (Other): patients with colonic adenomas who will undergo to laparoscopic segmental resection
  Interventions: Procedure: laparoscopic colon resection
- full-thickness laparo-endoscopic colon adenomas excision (Experimental): patients with colonic adenomas who will undergo to laparo-endoscopic full-thickness colon resection
  Interventions: Procedure: full-thickness laparo-endoscopic colon adenomas excision

INTERVENTIONS:
Procedure: full-thickness laparo-endoscopic colon adenomas excision — Full-thickness laparo-endoscopic removal of colon adenomas will be performed as follows: an endoscopist during intraoperative colonoscopy visualize the neoplasm, intra-luminary marks the margins of resection and stop at this in some cases. In another one: endoscopist start full-thickness removal of this lesion then the abdominal team during laparoscopy, with using laparoscopic technique, performe full-thickness resection of intestine wall with the tumor. Speciment extracted intralumenary or via minilaparotomy. Defect of the intestinal wall is sutured intracorporeally using laparoscopic technic. Desuflation, suturing of trocar sites.
  Arms: full-thickness laparo-endoscopic colon adenomas excision
Procedure: laparoscopic colon resection — Standard laparoscopic colon resection
  Arms: laparoscopic resection

SUMMARY:
Adenoma - carcinoma is a classic pathway of carcinogenesis. On this basis, timely removal of colon adenomas is a prophylactic measure to prevent colon cancer.

The standard treatment of colorectal adenomas is endoscopic mucosal resection or submucosal dissection (ESD). In 10 - 15% of cases the ESD is impossible, due to the size of the tumor, inconvenient localisation in the area of the diverticulum or appendix, the presence of fibrosis in the submucosal layer (Currie AC framework IDEAL // Colorectal Disease. 2019. No. 9 (21). P. 1004-1016.), (Suzuki S. Short-term results of laparoscopic endoscopic cooperative surgery of colorectal tumors (LECS-CR) in cases of endoscopically inoperable colorectal tumors // Surgery today . 2019. No. 12 (49). S. 1051-1057.). In that cases the segmental colectomy is justified.

An alternative to colectomy is a hybrid laparo-endoscopic surgery, which reduce postoperative hospital stay, incidence of complications and provide a comparable level of radicality (Lee SW, Garrett KA, Milsom JW Combined endoscopic and laparoscopic surgery (CELS) // Seminars on surgery of the colon and rectum. 2017. No. 1 (28). S. 24-29).

Thus, the planned study will contribute to the introduction into practice of an alternative method of management with tumors of the colon without signs of invasive growth when the endoscopically removal is impossible.

DETAILED DESCRIPTION:
During the study we will recruit the patients with colon epithelial tumors without signs of invasive growth which that cannot be removed endoscopically. In case of high risk of conversion endoscopic procedure the patient will be discussed on MD consillium. All of them will be informed about the possibility of resection methods in the absence of using endoscopic technics. Then the patients will be prepared for the operation in accordance with the method adopted in the clinic. At first colonoscopy will be performed in the operating room. Those patients for whom to perform endoscopic removal of the formation is impossible will be randomized intraoperatively using an Internet resource into 2 groups (main and comparison group).

The patients of the main group will undergo to hybrid laparo-endoscopic operation and comparative group - to laparoscopic colon resection.

After surgical procedure a pathomorphological examination of the speciments will performed with assessment of its quality. Postoperative complications in both groups will be recorded in accordance with the Clavien-Dindo classification. The level of postoperative pain will also be registred according to the visual analogue pain scale (VAS). Also we will be study the time of activation of patients, patient self-care scope according to the Bartell scale, postoperative hospital stay will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age is 18 years and older
2. Patients with colonic epithelial neoplasms without signs of invasive growth and not removable endoscopically
3. Informed agreement

Exclusion Criteria:

1. Positive regional lymph nodes
2. FAP
3. The presence of an intestinal stoma
4. ASI > III
5. Patients with IBD
6. Refusal of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
R1 resection rate | 30 days
  In according to pathological examination

SECONDARY OUTCOMES:
The level of postoperative pain | 10 days
  The level of postoperative pain with using a visual analogue pain scale: The patient assesses the postoperative pain from 0 to 10 points (0 points - no pain, 10 - unbearable pain).
The incidence and structure of postoperative complications | 30 days
  The incidence and structure of postoperative complications according to the Clavien-Dindo scale (I-grade - any deviation from the normal course of the postoperative course without the need for pharmacological, surgical, endoscopic or interventional radiological interventions. drugs that are acceptable include antiemetics, antipyretics, analgesics, diuretics, and electrolytes. In addition, this grade includes a wound infection "stopped at the patient's bedside", V grades - Death of the patient)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksey Kolosov, Study Chair — Ryzhikh National Medical Research Center of Coloproctology, Moscow, Russian Federation
Locations (1):
- Ryzhikh National Medical Research Center of Coloproctology, Moscow, Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No